CLINICAL TRIAL: NCT05577078
Title: TriBEL Registry: National Belgian Registry of Percutaneous Tricuspid Valve Repair Using a Transcatheter Edge-to-edge Repair Technique
Acronym: TriBEL
Status: Not yet recruiting | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Van der Heyden, Principal Investigator, AZ Sint-Jan AV
Other Study IDs: TriBEL
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Tricuspid Valve Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TEER: Patients with tricuspid valve regurgitation eligible for transcatheter edge-to-edge repair (TEER)
  Interventions: Procedure: Transcatheter edge-to-edge repair (TEER)

INTERVENTIONS:
Procedure: Transcatheter edge-to-edge repair (TEER) — Minimally invasive transcatheter-based edge-to-edge repair technique for tricuspid regurgitation

SUMMARY:
In this study, patients who have undergone or will undergo a transcatheter edge-to-edge repair (TEER) for tricuspid valve regurgitation (TR) will be followed up for 5 years. The goal of this prospective and retrospective, observational, non-randomized, multicenter registry is to confirm that TEER is a feasible, safe and effective treatment option for TR and to evaluate the long-term efficacy and safety of TEER.

The main endpoints are:

* Change in tricuspid regurgitation grade: number of patients with a reduction in tricuspid regurgitation score by at least one grade
* Composite of major adverse event: number of patients with composite of major adverse event (cardiovascular mortality, acute kidney injury, myocardial infarction, stroke or TIA, coronary revascularization, new onset AF or ventricular arrhythmia)

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Eligible for TEER procedure
* Informed consent signed

Exclusion Criteria:

* Unwilling to provide informed consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tricuspid valve regurgitation eligible for transcatheter edge-to-edge repair
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a reduction in tricuspid regurgitation score by at least one grade | 30 days
  Number of patients with a reduction in tricuspid regurgitation score by at least one grade 30 days post-procedure
Composite of major adverse event | 1 year
  Number of patients with composite of major adverse event (cardiovascular mortality, acute kidney injury, myocardial infarction, stroke or TIA, coronary revascularization, new onset AF or ventricular arrhythmia)

SECONDARY OUTCOMES:
Number of patients with a reduction in tricuspid regurgitation score by at least one grade at 6 months post-procedure | 6 months
  Number of patients with a reduction in tricuspid regurgitation score by at least one grade 6 months post-procedure
Number of patients with a reduction in tricuspid regurgitation score by at least one grade 1 year post-procedure | 1 year
  Number of patients with a reduction in tricuspid regurgitation score by at least one grade 1 year post-procedure
Number of patients with a reduction in tricuspid regurgitation score by at least one grade 2 years post-procedure | 2 years
  Number of patients with a reduction in tricuspid regurgitation score by at least one grade 2 years post-procedure
Number of patients with a reduction in tricuspid regurgitation score by at least one grade 3 years post-procedure | 3 years
  Number of patients with a reduction in tricuspid regurgitation score by at least one grade 3 years post-procedure
Number of patients with a reduction in tricuspid regurgitation score by at least one grade 4 years post-procedure | 4 years
  Number of patients with a reduction in tricuspid regurgitation score by at least one grade 4 years post-procedure
Number of patients with a reduction in tricuspid regurgitation score by at least one grade 5 years post-procedure | 5 years
  Number of patients with a reduction in tricuspid regurgitation score by at least one grade 5 years post-procedure
Composite of major adverse event at discharge | 5 days
  Number of patients with composite of major adverse event (cardiovascular mortality, acute kidney injury, myocardial infarction, stroke or TIA, coronary revascularization, new onset AF or ventricular arrhythmia) at discharge
Composite of major adverse event at 5 years post-procedure | 5 years
  Number of patients with composite of major adverse event (cardiovascular mortality, acute kidney injury, myocardial infarction, stroke or TIA, coronary revascularization, new onset AF or ventricular arrhythmia) 5 years post-procedure